CLINICAL TRIAL: NCT01934049
Title: The Effect of Dexmedetomidine on Postoperative Recovery in Elderly Patients With Femoral Neck Fracture Undergoing Hip Hemi-arthroplasty
Brief Title: Postoperative Recovery in Elderly Patients Undergoing Hip Hemi-arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Junle Liu, Principal Investigator, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dex-THR
Record Dates: First submitted 2013-08-21; First posted 2013-09-04 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Femoral Neck Fractures; Postoperative Complications; Inflammatory Response; Postoperative Delirium; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Femoral Neck Fractures; Postoperative Complications; Emergence Delirium; Postoperative Cognitive Complications | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Active Comparator): Dexmedetomidine in dex group is administered as 1ug/kg by intravenous infusion 10 min and then 0.6 ug/kg until 30 minutes before the operation finishes.
  Interventions: Procedure: hip arthroplasty; Drug: Total Intravenous Anesthesia and Peripheral nerve blocks
- Saline (Placebo Comparator): Participants in con group receive placebo(saline) as the same dose at the same time as dex group.
  Interventions: Procedure: hip arthroplasty; Drug: Total Intravenous Anesthesia and Peripheral nerve blocks

INTERVENTIONS:
Procedure: hip arthroplasty — Every patient with femoral neck fractures must undergo hip hemi-arthroplasty.
Drug: Total Intravenous Anesthesia and Peripheral nerve blocks — Every patient receives Peripheral nerve blocks and Total Intravenous Anesthesia with propofol

SUMMARY:
Hip fractures incidence grows rapidly with the aging of the population. After indicated surgical treatment, hip fracture patients experience high rates of postoperative complications, postoperative delirium (PD), postoperative cognitive dysfunction (POCD), leading to poor postoperative recovery during hospitalization, which can cause disability, distress for both patients and their families, are associated with other medical complications and account for significant additional health care costs. We currently use dexmedetomidine in elderly patients with hip fractures undergoing hip hemi-arthroplasty in order to improve postoperative recovery and prevent and treating PD and POCD.

Dexmedetomidine is a drug used for sedation in critically ill patients that provides some pain relief and controls the bodies response to stress. The sedation produced by dexmedetomidine appears more similar to natural sleep than any other drug used for anesthesia and postoperative sedation. Data suggesting that dexmedetomidine can prevent delirium following cardiac surgery and the developing understanding of the causes of PD and POCD suggest that dexmedetomidine will be particularly effective.

ELIGIBILITY:
Inclusion criteria

* Age > 75years old
* Patients with femoral neck fractures
* Undergoing hip hemi-arthroplasty surgery
* American Society of Anesthesiologists (ASA) physical status II-IV
* MoCA being more than 23

Exclusion Criteria

* Patient refusal to participate in the study
* Patient refusal or failure of regional block
* allergic to local anesthetics or general anesthetics
* history of opioid dependence
* contraindications to nerve blocks (coagulation defects, infection at puncture site, preexisting neurological deficits in the lower extremities)
* current severe psychiatric disease or alcoholism or drug dependence
* severe visual or auditory disorder

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-02 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
postoperative cognitive dysfunction(POCD) | 7days
  POCD is assessed by Montreal Cognitive Assessment(MoCA), which was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration,executive functions, memory, language,visuoconstructional skills, conceptual thinking,calculations, and orientation. Time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points; a score of 26 or above is considered normal.

SECONDARY OUTCOMES:
Postoperative recovery | 7days
  The postoperative recovery is assessed by the Post-operative Quality Recovery Scale (PQRS),which is a research tool designed to measure postoperative quality of recovery in multiple domains and over multiple time periods. Recovery domains include physiological, emotive (depression and anxiety), nociceptive (pain and nausea), cognitive, activities of daily living (ADL), and overall patient perspective (including satisfaction).
Postoperative Delirium(PD) | 72 hours
  The postoperative Delirium is assessed by the Confusion Assessment Method (CAM)

OTHER OUTCOMES:
postoperative complications | 7 days
perioperative opioid consumption | 3 days
  Intraoperative and postoperative opioid consumption were calculated between the two groups.
IL-6 and C-reacting protein | 7 days
MB isoenzyme of creatine kinase and blood sugar | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: zhang hong, ph.d, Study Chair — Anesthesia and Operation Center, Chinese People's Liberation Army General Hospital
Locations (1):
- Anesthesia and Operation Center, Chinese People's Liberation Army General Hospital, Beijing, China